CLINICAL TRIAL: NCT00671073
Title: Phase II Dose-Ranging Study of the Efficacy and Safety of Oglemilast in Patients With COPD
Brief Title: Study To Assess Efficacy and Safety of Oglemilast in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRC-MD-50
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Pulmonary Disease; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; COPD; COAD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — oglemilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Oglemilast low dose, oral administration once daily for 12 weeks
  Interventions: Drug: Oglemilast
- 2 (Active Comparator): Oglemilast middle dose, oral administration, once daily for 12 weeks
  Interventions: Drug: Oglemilast
- 3 (Active Comparator): Oglemilast high dose, oral administration, once daily for 12 weeks.
  Interventions: Drug: Oglemilast
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oglemilast — Oglemilast low dose, oral administration, once daily for 12 weeks
  Other Names: GRC 3886
  Arms: 1
Drug: Placebo — Placebo, oral administration, once daily for 12 weeks
  Arms: 4
Drug: Oglemilast — Oglemilast middle dose, oral administration, once daily for 12 weeks
  Other Names: GRC 3886
  Arms: 2
Drug: Oglemilast — Oglemilast high dose, oral administration, once daily for 12 weeks
  Other Names: GRC 3886
  Arms: 3

SUMMARY:
This study will assess the safety and efficacy of a range of oglemilast doses. The study will be 14 weeks in duration. All patients meeting the eligibility criteria will be randomized to one of three doses of oglemilast or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Presence of COPD as defined by GOLD criteria (2006); post-bronchodilator FEV1/FVC <70%, and post-bronchodilator FEV1 >30% and < 80% predicted
* Current or former cigarette smoker

Exclusion Criteria:

* Long-term oxygen use of > 15 hours a day
* Symptoms consistent with a significant asthmatic component (e.g. atopic disease, allergic symptoms)
* Any COPD exacerbations within 30 days prior to study entry or during run-in
* History of chronic or recurrent gastrointestinal disorder associated with bleeding in previous 12 months
* Presence of clinical significant pulmonary disease other than COPD

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2008-05-05; Primary Completion 2009-05-15 (Actual); Study Completion 2009-05-15 (Actual)

PRIMARY OUTCOMES:
Pre-bronchodilator morning (trough) forced expiratory volume in 1 second (FEV1) | After 12 weeks of treatment

SECONDARY OUTCOMES:
Pre-bronchodilator forced vital capacity (FVC) | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Maurer, MS, Study Director — Forest Laboratories
Locations (44):
- United States (44):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Tucson, Arizona
  - Forest Investigative Site, Buena Park, California
  - Forest Investigative Site, Encinitas, California
  - Forest Investigative Site, Fullerton, California
  - Forest Investigative Site, Los Angeles, California
  - Forest Investigative Site, Orange, California
  - Forest Investigative Site, Rancho Mirage, California
  - Forest Investigative Site, San Diego, California
  - Forest Investigative Site, Stockton, California
  - Forest Investigative Site, Centennial, Colorado
  - Forest Investigative Site WR1, Wheat Ridge, Colorado
  - Forest Investigative Site WR2, Wheat Ridge, Colorado
  - Forest Investigative Site, Waterbury, Connecticut
  - Forest Investigative Site, Fort Lauderdale, Florida
  - Forest Investigative Site, Miami, Florida
  - Forest Investigative Site, Ormond Beach, Florida
  - Forest Investigative Site, Tamarac, Florida
  - Forest Investigative Site, Skokie, Illinois
  - Forest Investigative Site, Evansville, Indiana
  - Forest Investigative Site, North Dartmouth, Massachusetts
  - Forest Investigative Site, Livonia, Michigan
  - Forest Investigative Site, Edina, Minnesota
  - Forest Investigative Site, Minneapolis, Minnesota
  - Forest Investigative Site, Papillion, Nebraska
  - Forest Investigative Site, Cherry Hill, New Jersey
  - Forest Investigative Site, Elmira, New York
  - Forest Investigative Site, Mineola, New York
  - Forest Investigative Site, Rochester, New York
  - Forest Investigative Site, Charlotte, North Carolina
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Toledo, Ohio
  - Forest Investigative Site, Medford, Oregon
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Bethlehem, Pennsylvania
  - Forest Investigative Site, Philadelphia, Pennsylvania
  - Forest Investigative Site, Charleston, South Carolina
  - Forest Investigative Site, Greenville, South Carolina
  - Forest Investigative Site, Spartanburg, South Carolina
  - Forest Investigative Site, El Paso, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Fredericksburg, Virginia
  - Forest Investigative Site, Tacoma, Washington